CLINICAL TRIAL: NCT01250717
Title: Docetaxel Followed by Radical Prostatectomy in Patients With High Risk Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Glenn Bubley, MD, Director Of Genitourinary Oncology @ Beth Israel Deaconess Medical Center, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001P-001577; E-99-0363-FB (Other: BIDMC IRB)
Record Dates: First submitted 2010-11-23; First posted 2010-12-01 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2012-08

CONDITIONS: Prostate Cancer
Keywords: prostatectomy; docetaxel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Dexamethasone; Calcium Dobesilate; Estramustine; Goserelin; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel Followed by Radical Prostatectomy (Experimental): Docetaxel,Dexamethasone,Estramustine,Zoladex,Casodex,Prostatectomy
  Interventions: Drug: Docetaxel; Drug: Dexamethasone; Drug: Estramustine; Drug: Zoladex; Drug: Casodex; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Docetaxel — Given by an IV infusion over 1 hour on day 2 of a three-week cycle
  Other Names: Taxotere
Drug: Dexamethasone — Orally 12 hours and 1 hour before docetaxel and again 12 hours after docetaxel
  Other Names: Decadron
Drug: Estramustine — Taken orally three times a day for 5 days for the first part of every three week cycle
Drug: Zoladex — Given subcutaneously for 4 doses every three months
  Other Names: goserelin acetate
Drug: Casodex — Taken orally once a day for 6 months
  Other Names: Bicalutamide
Procedure: Radical Prostatectomy — after the chemo and hormonal therapy all patients have a radiacal prostatectomy

SUMMARY:
The purpose of this research study is to determine if the combination of chemotherapy and hormone therapy is safe and helpful for patients who plan to have their high-risk prostate cancer surgically removed. Some physicians believe that patients with high risk cancer that is located in one area, may have an early but small spread of the cancer outside of the prostate, and perhaps even to distant organs. Therefore, better treatments for the entire body are needed to improve the ability of surgery or other local therapies to cure prostate cancer. Since chemotherapy is beginning to demonstrate increasing activity in advanced prostate cancer patients, it is possible that using chemotherapy combined with hormonal therapy earlier in the course of localized but high risk patients might improve the outcomes for these patients.

DETAILED DESCRIPTION:
* Participants will receive treatment in the outpatient clinic, where the docetaxel chemotherapy will be placed in a bag of fluid and will be given by vein every three weeks. Participants will take Decadron (dexamethasone) by mouth 12 hours and 1 hour before docetaxel and again 12 hours after docetaxel. They will also take estramustine and casodex by mouth at home. Zoladex (or lupron) will be given subcutaneously (under the skin) 4 times every three months. They will also be started on coumadin beginning at the time of the first docetaxel infusion and continuing until 3 weeks after the 4th cycle of chemotherapy.
* After 2 months (or cycles) of therapy, participants will be evaluated in order to assess the response and toxicity of treatment, including a review of medical history, physical examination, blood tests, including PSA. If there is no evidence of progression or excessive toxicity, treatment will continue for 2 more months in the same manner.
* At the end of 4 months of chemotherapy, participants will be reassessed by the medical oncologist and urologist regarding surgery to remove the prostate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Potential candidate for radical prostatectomy
* Any of the following: a) clinical stage T3 patients, b) Serum PSA greater than or equal to 20 ng/ml, c) Gleason score 8-10, d) Clinical T2 disease and either MRI evidence of seminal vesicle involvement or Gleason 4+3 cancer with either 5 or 6 biopsies positive
* ECOG Performance Status 0-1
* WBC > 3,000 ul
* HCT > 30%
* PLT > 100,000/ul
* LFTS within normal limits

Exclusion Criteria:

* Prior hormones, radiation or chemotherapy for prostate cancer
* Myocardial infarction within 1 year, significant change in anginal pattern within last 6 months, current congestive heart failure (NYHA Class 2 or higher), or deep venous thrombosis within 1 year
* Evidence of active infection
* Significant peripheral neuropathy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2001-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J. Bubley, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 28, 1999 and May 17, 2005, 28 participants with high risk localized prostate cancer were enrolled on this IRB approved phase II protocol from BIDMC Urology clinics
Pre-assignment Details: This was a single arm study and there were no arms. Participants were screened for final eligibility after consent was completed. All enrolled subjects were treated
Groups:
- Docetaxel Followed by Radical Prostatectomy: This is a single arm study and there were no arms other than the one arm. All participants were treated according to the regimen below.
  Docetaxel Followed by Radical Prostatectomy
  Radical Prostatectomy : after the chemo and hormonal therapy all patients have a radical prostatectomy
  Zoladex : Given subcutaneously for 4 doses every three months
  Casodex : Taken orally once a day for 6 months
  Estramustine : Taken orally three times a day for 5 days for the first part of every three week cycle
  Docetaxel : Given by an IV infusion over 1 hour on day 2 of a three-week cycle
  Dexamethasone : Orally 12 hours and 1 hour before docetaxel and again 12 hours after docetaxel
Period: Overall Study
Arm/Group | Docetaxel Followed by Radical Prostatectomy
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel Followed by Radical Prostatectomy
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 57 (NA) [43 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Was Assessed by Rigorous Pathological Examination by One of Two Pathologists
Description: One of two pathologists (SR, EG), assigned the Gleason scores for each patient from pre-treatment prostate biopsies and assessed pathological staging on post- prostatectomy specimens. Staging including a description of all tumor foci within the gland, presence or absence of perineural invasion and/or lymphovascular invasion, presence of extraprostatic extension of tumor (including seminal vesicle invasion), and margin status. The pathologists reviewed the presence or absence of cancer in each prostate gland removed on the study patients. RECIST has to my knowledge not been used for pathological examination in neoadjuvant studies. 0 out of 28 participants acheived complete response. RECIST is not appropriate as cancer within the gland at the time of treatment is not measurable by RECIST. The primary outcome is a pathological complete response.
Time Frame: status post prostectomy
Measure: Number; unit: participants
Arm/Group | Docetaxel Followed by Radical Prostatectomy
Number analyzed (Participants) | 28
participants | 0
Statistical Analysis 1: Comparison: Docetaxel Followed by Radical Prostatectomy; Test type: Superiority or Other; Percentage = 0, 95% CI 2-sided [0 to 0.12]

ADVERSE EVENTS:
Time Frame: 6 months
Description: followed for four cycles of therapy
Arm/Group | Docetaxel Followed by Radical Prostatectomy
Serious Adverse Events (participants affected / at risk) | 5/28
Other Adverse Events (participants affected / at risk) | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel Followed by Radical Prostatectomy (N=28)
neutropenic fever (Blood and lymphatic system disorders) | 4 (4) — defined as ANC < 500 and fever over 100 degrees farenheit
elevated liver functions (Hepatobiliary disorders) | 1 (1) — assessment by ALT and AST levels with 3.0 common toxicity criteria

LIMITATIONS AND CAVEATS:
Although this study has the longest median follow-up periods reported (80 months or 6.6 years), the overall number of participants is too few to make strong judgements about efficacy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No